CLINICAL TRIAL: NCT06353737
Title: Looking for Asymptomatic Mpox in a Population at High Risk
Acronym: LAMP
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: CTO 4489
Record Dates: First submitted 2024-04-02; First posted 2024-04-09 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Mpox (Monkeypox)
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mpox is caused by a virus that can be spread through touching the affected skin of someone who has the infection, touching sheets or clothes that has been used by someone with the infection, or breathing in particles of virus from someone who has the infection. Mpox infection can cause skin and flu-like symptoms, but can also cause very few symptoms, or no symptoms at all. While the number of participants with mpox symptoms can be tracked, little is known about how many people have mpox, but experience few or no symptoms at all. To do this, a Canadian sample of gay, bisexual and other men who have sex with men (GBMSM) who are participating in a randomized controlled trial will be screened for mpox symptoms. Screening will include questions about whether they may be experiencing any mpox symptoms, history of past diagnosis of mpox, sexual history, and vaccination history and awareness. Swabs will be taken to test for the presence of mpox virus, and a blood sample will be taken to test for antibodies. Approximately 450 individuals will be recruited. The results will be descriptive in nature.

ELIGIBILITY:
Inclusion criteria:

- Participants need to have been enrolled in an existing randomized clinical trial (NCT04762134)

Exclusion criteria:

- None

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Gay, bisexual, and other men who have sex with men
Study Population: Participants need to have been enrolled in an existing randomized clinical trial (NCT04762134)
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Asymptomatic prevalence | 2 weeks
  To determine the prevalence of asymptomatic, pre-symptomatic and paucisymptomatic mpox infection (pooled and individually), in a population of GBMSM with anticipated high mpox risk and high prevalence of vaccination.

SECONDARY OUTCOMES:
Symptomatic prevalence | 2 weeks
  To determine the prevalence of symptomatic mpox infection in the study sample
Mpox seropositivity | 2 weeks
  To determine the prevalence of mpox seropositivity (both for total antibody and for neutralizing antibody) in the study sample
Characteristics | 2 weeks
  To identify clinical and demographic characteristics associated with asymptomatic and/or paucisymptomatic infection in the study sample
Characteristics of seropositivity | 2 weeks
  To identify clinical and demographic characteristics associated with mpox seropositivity in the study sample

CONTACTS AND LOCATIONS:
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Group level data will be made available upon request